CLINICAL TRIAL: NCT04270045
Title: Forced Oscillometry in Infants With Bronchopulmonary Dysplasia
Status: Recruiting | Type: Observational
Sponsor: Winston Manimtim (Other)
Responsible Party: Sponsor-Investigator, Winston Manimtim, Principal Investigator, Children's Mercy Hospital Kansas City
Organization: Children's Mercy Hospital Kansas City (Other)
Other Study IDs: STUDY00000912
Record Dates: First submitted 2020-02-11; First posted 2020-02-17 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Infant, Premature, Diseases; Bronchopulmonary Dysplasia; Respiratory Distress Syndrome
MeSH Terms: conditions — Infant, Premature, Diseases; Bronchopulmonary Dysplasia; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single: Non-invasive forced airway oscillometry. Normative data will be established form term neonates without pulmonary disease
  Interventions: Device: Non-invasive forced airway oscillometry

INTERVENTIONS:
Device: Non-invasive forced airway oscillometry — This non-invasive device will measure pulmonary mechanics in spontaneously breathing premature infants and term infants without pulmonary disease. Infant will be in supine position and breathing regularly. A cushioned mask will be placed on the infant's face, covering the nose and mouth. Measurements typically take less than 20 seconds and no more than 3 repetitions will be done at each time point.

SUMMARY:
The purpose of this study is to use forced oscillometry technique (FOT) to measure pulmonary mechanics and function in in term infants and premature infants with bronchopulmonary dysplasia (BPD)

DETAILED DESCRIPTION:
Pulmonary function testing has been the standard of care to diagnose and evaluate response to therapy in various respiratory diseases in adults and children. There are several equipment and techniques that are FDA approved for these purposes. However, there are currently no lung function tests that are practically feasible, clinically meaningful and widely used in infants.

The forced oscillation technique (FOT) is a non-invasive method that had been used to measure respiratory mechanics. FOT employs small amplitude pressure oscillations superimposed on the normal breathing and therefore has the advantage over conventional lung function techniques that it does not require the performance of respiratory maneuvers. To date, the use of this technique is FDA approved in adults and children but remains largely experimental in infants and newborns. THORASYS has recently developed a new respiratory function test device aimed specifically at newborn and infants (0 - 2 years age group) called tremoflo N-100 ("Neo"). This new device measures lung function in only a few minutes while the newborn or infant is sleeping normally. It uses an adapted version of the Airwave Oscillometry (AOS) to calculate the impedance of the lungs and quantify airway obstruction.

Diuretics and bronchodilators are two on the most commonly used medications to ameliorate the symptoms of BPD. The benefits of these therapies have not been shown to prevent the development of BPD in a randomized control trial (RCT). More recently, there have been some evidence from pharmacogenetic studies that the variability in bronchodilator responsiveness in patients with asthma, (and possibly BPD) may lie on the gene encoding the B2-adrenergic receptor (ADRB2) as well as within the associated G-protein receptor pathway, the nitric oxide biosynthetic pathway and other novel loci identified in recent genome-wide studies. This part of the study will be hypothesis generating to try to understand the variability in bronchodilator response in infants with BPD. Normative data will be established in term neonates.

ELIGIBILITY:
Inclusion Criteria:

Preterm Cohort:

* Premature infants with BPD who are in room air based on the (per NICHD definition)
* Premature infants with BPD who are receiving low flow O2 support and able to maintain normal spO2 in Room air for brief period ( up to 3 minutes) Term Cohort without pulmonary disease
* Infants >36 weeks gestational age without pulmonary disease
* Infants < 4 weeks of age

Outpatient Cohort:

* Former preterm infants < 32 weeks at birth
* Those with BPD based on NIH 2001 definition
* Seen prior to 2 years of age

Exclusion Criteria:

* Infants with BPD requiring invasive or non-invasive positive pressure ventilation
* Infants with BPD who have associated genetic diagnosis or major congenital anomalies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Premature infants with bronchopulmonary Dysplasia who are in room air or Premature infants with BPD who are receiving low flow O2 support and able to maintain normal spO2 in Room air for brief period (up to 3 minutes) Term infants without pulmonary disease. Former preterm infants (<32 weeks) with BPD seen prior to 2 years of age in the outpatient setting.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-02-06 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Forced oscillation technique measurements | FOT measurement prior to bronchodilator therapy
  Baseline FOT measurements in premature infants with BPD and term infants without pulmonary disease.
Post-bronchodilator forced oscillation technique measurements (in subjects already receiving this therapy) | FOT measurement 30 to 60minutes following bronchodilator therapy
  FOT measurements in premature infants with BPD following bronchodilator therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No